CLINICAL TRIAL: NCT00680368
Title: Resident Supervision Index: Assessing Feasibility and Validity
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: SHP 08-164
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2014-12-16 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Feasibility; Supervision; Assessing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — The study did not involve a biospecimen. None was collected. None was retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Residents and Attending Physicians: This group contains the residents and the attending physicians who consented to participate in the study. They participated in a survey administered by a research assistant. Both physician resident and attending physicians were administered the survey twice within 24-hours and their test-retest responses were compared for reliability. Responses to attending and resident physicians covering the care for the patient and clinical care encounter were compared for accuracy.

SUMMARY:
OBJECTIVES: To develop, assess feasibility, and test the validity of the Resident Supervision Index (RSI), a survey tool for medical residents designed to measure quantitatively the level of supervision the resident received while caring for an outpatient during a patient care encounter.

RESEARCH DESIGN: This is a prospective trial assessing the Residency Supervision Index (Index) applied to outpatient care encounters for content validity, test-retest reliability, and construct validity.

DETAILED DESCRIPTION:
OBJECTIVES: To develop, assess feasibility, and test the validity of the Resident Supervision Index (RSI), a survey tool for medical residents designed to measure quantitatively the level of supervision the resident received while caring for an outpatient during a patient care encounter.

RESEARCH DESIGN: This is a prospective trial assessing the Residency Supervision Index (Index) applied to outpatient care encounters for test-retest reliability and construct validity.

METHODOLOGY: Trained interviewers administered the Index during face-to-face and in-clinic interviews with 60 consenting resident physicians and their 37 consenting attending physicians to descsribe the care they provided to 143 patients at the outpatient clinics involving 148 clinical encounters at the Loma Linda VA Medical Center.

For each encounter, data comes from administering the Resident Supervision Index to the resident and attending. Baseline data describing each subject (attending physicians and resident physicians) came from face-to-face interviews.

Test-retest reliability is assessed by re-administering the Index to residents for within 24 hours of the encounter. Concurrent validity is assessed by re-administering the Index to the attending physician responsible for the patient's care.

CLINICAL RELATIONSHIPS: The study will help our understanding of how residents at VA medical centers receive training and are supervised for the purpose of both education and patient outcomes.

IMPACT/SIGNIFICANCE: The instrument is planned for future studies to assess the association between resident supervision and training outcomes, clinical workload, patient outcomes, quality of care, and care costs.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Ages 18 and older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrell Michael Kashner, PhD JD MPH, Principal Investigator — VA Loma Linda Healthcare System, Loma Linda, CA; Dale S. Cannon, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California, United States

REFERENCES:
- [Background] Cannon GW, Keitz SA, Holland GJ, Chang BK, Byrne JM, Tomolo A, Aron DC, Wicker AB, Kashner TM. Factors determining medical students' and residents' satisfaction during VA-based training: findings from the VA Learners' Perceptions Survey. Acad Med. 2008 Jun;83(6):611-20. doi: 10.1097/ACM.0b013e3181722e97. PMID 18520472
- [Background] Kashner TM, Henley SS, Golden RM, Byrne JM, Keitz SA, Cannon GW, Chang BK, Holland GJ, Aron DC, Muchmore EA, Wicker A, White H. Studying the effects of ACGME duty hours limits on resident satisfaction: results from VA learners' perceptions survey. Acad Med. 2010 Jul;85(7):1130-9. doi: 10.1097/ACM.0b013e3181e1d7e3. PMID 20592508
- [Result] Byrne JM, Kashner M, Gilman SC, Aron DC, Cannon GW, Chang BK, Godleski L, Golden RM, Henley SS, Holland GJ, Kaminetzky CP, Keitz SA, Kirsh S, Muchmore EA, Wicker AB. Measuring the intensity of resident supervision in the department of veterans affairs: the resident supervision index. Acad Med. 2010 Jul;85(7):1171-81. doi: 10.1097/ACM.0b013e3181d5a954. PMID 20305532
- [Result] Kashner TM, Byrne JM, Henley SS, Golden RM, Aron DC, Cannon GW, Chang BK, Gilman SC, Holland GJ, Kaminetzky CP, Keitz SA, Muchmore EA, Kashner TK, Wicker AB. Measuring progressive independence with the resident supervision index: theoretical approach. J Grad Med Educ. 2010 Mar;2(1):8-16. doi: 10.4300/JGME-D-09-00083.1. PMID 21975879
- [Result] Kashner TM, Byrne JM, Chang BK, Henley SS, Golden RM, Aron DC, Cannon GW, Gilman SC, Holland GJ, Kaminetzky CP, Keitz SA, Muchmore EA, Kashner TK, Wicker AB. Measuring progressive independence with the resident supervision index: empirical approach. J Grad Med Educ. 2010 Mar;2(1):17-30. doi: 10.4300/1949-8357-2.1.17. PMID 21975880

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: The study began with 112 responders: 75 physician residents and 37 attending physicians. Only 60 of the 75 residents had been supervised by one of the 37 participating attending physicians. Thus, 15 residents were dropped from study. Both resident and their attending physician were surveyed to report total supervision time for each of 148 clinical encounters with 143 patients. There were more clinical encounters than patients because some patients had more than one encounter. There were more physician residents than attending physicians because attending physicians may have supervised more than one resident. There were more clinical encounters than residents because a resident may be involved in more than one clinical encounter with a patient.
Period: Overall Study
Arm/Group | Group 1
Started | 112
Completed | 97 (15 residents excluded because their attending physician was not participating in the study)
Not Completed | 15
Not completed — not supervised, not eligible | 15

BASELINE CHARACTERISTICS:
Population: Physician residents who consented to participate in the study.
Groups:
- Physician Residents and Attending Physicians: includes physician residents and attending physicians who were asked to sit through a face to face interview with a research assistant following a clinical encounter with a patient
Arm/Group | Physician Residents and Attending Physicians
Number analyzed (Participants) | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 112
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 72

OUTCOME MEASURES:

1. Primary Outcome: Intraclass Correlation Coefficient Between Physician Resident and Attending Physician.
Description: Describes agreement between physician resident and attending physician assessment of total resident supervision time for a given patient and patient care clinical encounter.
Time Frame: 24-hours
Measure: Number (95% Confidence Interval); unit: Intraclass Correlation Coefficient
Groups:
- Physician Residents and Attending Physicians: Sample included 112, including 60 physician residents and 37 attending physicians
Arm/Group | Physician Residents and Attending Physicians
Number analyzed (Participants) | 97
Intraclass Correlation Coefficient | .69 [.57 to .78]

2. Secondary Outcome: Intraclass Correlation Coefficient Assessing Test-retest Reliability for Resident Physicians
Description: Assesses the test-retest reliability of repeated responses for resident physicians only to report the total time spent during resident supervision.
Time Frame: 24 hours
Measure: Number (95% Confidence Interval); unit: Intraclass Correlation Coefficient
Groups:
- Physician Residents: Includes physician residents who had a supervising attending physician participating in the study, and who received a face to face interview with a research assistant
Arm/Group | Physician Residents
Number analyzed (Participants) | 60
Intraclass Correlation Coefficient | .93 [.91 to .95]

3. Secondary Outcome: Intraclass Correlation Coefficient for Test-retest Reliability for Attending Physicians
Description: Assesses the test-retest reliability among repeated responses to surveys administered to attending physicians only.
Time Frame: 24 hours
Measure: Number (95% Confidence Interval); unit: Intraclass Correlation Coefficient
Groups:
- Attending Physicians: Results reported only for the 37 attending physicians in the study sample
Arm/Group | Attending Physicians
Number analyzed (Participants) | 37
Intraclass Correlation Coefficient | .88 [.82 to .91]

ADVERSE EVENTS:
Time Frame: Collected during the 3-months when subjects were interviewed only.
Groups:
- Group 1: Sample included 75 resident physicians. No adverse events noted.
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=75)
quality of care (General disorders) | 0 (0) — There were no adverse health events.
Mental breakdown (Psychiatric disorders) | 0 (0) — Potential for mental breakdown due to stress of completing a survey in clinic
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=75)
dissatisfaction with education experience (General disorders) | 0 (0) — Reflects dissatisfaction with education experience
Eye strain (Eye disorders) | 0 (0) — Eye strain attempting to complete a survey

LIMITATIONS AND CAVEATS:
Single site study limiting generalizability of findings

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes